CLINICAL TRIAL: NCT06655558
Title: Validating the Clinical Effect of a Knee Orthosis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Budget for the research project ran out.
Sponsor: TOPMED (Other)
Collaborators: Natural Sciences and Engineering Research Council, Canada (Other); O3D inc. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 241_O3D_Quest
Record Dates: First submitted 2024-10-21; First posted 2024-10-23 (Actual); Results first posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Medial Gonarthrosis
Keywords: knee orthosis; knee brace; validation; WOMAC; knee pain; knee stiffness; daily activities; knee function

STUDY DESIGN:
Intervention Model Description: Longitudal treatment validation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- medial gonarthrosis (Experimental): Patients with medial gonarthrosis
  Interventions: Device: custom knee orthosis

INTERVENTIONS:
Device: custom knee orthosis — The custom knee orthosis will be worn for 8 weeks (56 days).

SUMMARY:
The aging population is steadily increasing, partly due to increasing life expectancy. At the same time, chronic diseases, including those affecting the musculoskeletal system (e.g., osteoarthritis), whose prevalence increases with age, limit the daily activities of those affected and thus affect more and more people. Arthrosis is the most common form of these diseases worldwide. According to the l'Institut de la statistique du Québec, nearly one in two Quebecers aged 15 and over is affected by a chronic health problem.

Knee orthosis is one form of treatment that helps patients suffering from knee gonarthrosis. This treatment aims to compensate for certain biomechanical deficits in patients. A variety of joint configurations exists to target specific biomechanical deficits. A constant challenge for companies manufacturing orthoses is transmitting the orthosis's biomechanical effect to the patient. The desired effect requires a change in the forces applied inside the knee, but the orthosis cannot directly transmit forces to the patient's bones due to its external nature to the body. Customization of orthoses is crucial to improve the transmission of the biomechanical effect as well as tolerance to it. O3D Inc. aims to validate the effectiveness of its new custom orthosis for treating knee gonarthrosis symptoms.

Participants answered a Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) questionnaire before receiving their custom knee brace(Baseline) and after 8 weeks (56 days) of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Suffering from medial gonarthrosis
* Receiving a regular model of the O3D orthosis

Exclusion Criteria:

* Suffering from tricompartmental gonarthosis
* Having completed the delivery appointment for a O3D orthosis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2024-07-31 (Actual); Primary Completion 2024-12-22 (Actual); Study Completion 2025-06-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edith Martin, Phd., Principal Investigator — TOPMED
Locations (1):
- Topmed, Québec, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Medial Gonarthrosis: Patients with medial gonarthrosis
  custom knee orthosis: The custom knee orthosis will be worn for 8 weeks.
Period: Overall Study
Arm/Group | Medial Gonarthrosis
Started | 2 (Participants with medial gonarthosis)
Completed | 1 (Participants with medial gonarthosis)
Not Completed | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Population: All participants who completed the study.
Arm/Group | Medial Gonarthrosis
Number analyzed (Participants) | 1
Age, Customized [Count of Participants; unit: Participants] — Participants aged between 18 and 75 years old inclusively.
  Participants
    18<age<75 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 1
WOMAC Total Score [Mean (Standard Deviation); unit: units on a scale] — Western Ontario and McMaster Universities Osteoarthritis Index(WOMAC) 24 item questionnaire about knee pain, stiffness and function. Each item uses a 5 point scale ranging from 0 (no pain, stiffness or difficulty) to 4 (extreme pain, stiffness or difficulty). Total score is the sum of all items and ranges from 0 to 96. Therefore low scores represent better knee health whereas high scores represent worse knee health.
  units on a scale | 52 (0)
WOMAC Pain score [Mean (Standard Deviation); unit: units on a scale] — Western Ontario and McMaster Universities Osteoarthritis Index(WOMAC) subcore of 5 items about knee pain. Each item uses a 5 point scale ranging from 0 (no pain) to 4 (extreme pain). Pain score is the sum of all 5 items, ranges from 0 to 20. Therefore low scores represent better knee pain whereas high scores represent worse knee pain.
  units on a scale | 10 (0)
WOMAC Stiffness Score [Mean (Standard Deviation); unit: units on a scale] — Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) subscore of 2 items about knee stiffness. Each item uses a 5 point scale ranging from 0 (no stiffness) to 4 (extreme stiffness). Stiffness score is the sum of 2 items, ranges from 0 to 8. Therefore low scores represent better knee stiffness whereas high scores represent worse knee stiffness.
  units on a scale | 5 (0)
WOMAC Physical Function Score [Mean (Standard Deviation); unit: units on a scale] — Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) subscore of 17 items about knee function. Each item uses a 5 point scale ranging from 0 (no dificulty) to 4 (extreme dificulty). Physical function score is the sum of all 17 items, ranges from 0 to 68. Therefore low scores represent better knee function whereas high scores represent worse knee function.
  units on a scale | 37 (0)

OUTCOME MEASURES:

1. Primary Outcome: Change in WOMAC Total Score
Description: Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) 24 item questionnaire about knee pain, stiffness and function. Each item uses a 5 point scale ranging from 0 (no pain, stiffness or difficulty) to 4 (extreme pain, stiffness or difficulty). Total score is the sum of all items and ranges from 0 to 96. Therefore low scores represent better knee health whereas high scores represent worse knee health. Change is calculated as :
  Change= Score after 8 weeks of treatment - Baseline Score
Time Frame: At baseline and after 8 weeks of intervention(Day 56)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Medial Gonarthrosis
Number analyzed (Participants) | 1
units on a scale | 6 (0)

2. Primary Outcome: Change in WOMAC Pain Score
Description: Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) subcore of 5 items about knee pain. Each item uses a 5 point scale ranging from 0 (no pain) to 4 (extreme pain). Pain score is the sum of all 5 items, ranges from 0 to 20. Therefore low scores represent better knee pain whereas high scores represent worse knee pain. Change is calculated as :
  Change= Score after 8 weeks of treatment - Baseline Score
Time Frame: At baseline and after 8 weeks of intervention(Day 56)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Medial Gonarthrosis
Number analyzed (Participants) | 1
units on a scale | 3 (0)

3. Primary Outcome: Change in WOMAC Stiffness Score
Description: Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) subscore of 2 items about knee stiffness. Each item uses a 5 point scale ranging from 0 (no stiffness) to 4 (extreme stiffness). Stiffness score is the sum of 2 items, ranges from 0 to 8. Therefore low scores represent better knee stiffness whereas high scores represent worse knee stiffness. Change is calculated as :
  Change= Score after 8 weeks of treatment - Baseline Score
Time Frame: At baseline and after 8 weeks of intervention(Day 56)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Medial Gonarthrosis
Number analyzed (Participants) | 1
units on a scale | 1 (0)

4. Primary Outcome: Change in WOMAC Physical Function Score
Description: Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) subscore of 17 items about knee function. Each item uses a 5 point scale ranging from 0 (no dificulty) to 4 (extreme dificulty). Functionnal limitation score is the sum of all 17 items, ranges from 0 to 68. Therefore low scores represent better knee function whereas high scores represent worse knee function. Change is calculated as :
  Change= Score after 8 weeks of treatment - Baseline Score
Time Frame: At baseline and after 8 weeks of intervention(Day 56)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Medial Gonarthrosis
Number analyzed (Participants) | 1
units on a scale | 2 (0)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected throughout the full duration of the protocol for each participant, therfore 8 weeks
Arm/Group | Medial Gonarthrosis
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

LIMITATIONS AND CAVEATS:
Targeted enrollement of 30 participants was not reached. Interpretations should be taken with caution because of the small number of participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is more than 60 days but less than or equal to 365 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2024-05-08): https://cdn.clinicaltrials.gov/large-docs/58/NCT06655558/Prot_000.pdf
  • Informed Consent Form (2024-05-08): https://cdn.clinicaltrials.gov/large-docs/58/NCT06655558/ICF_001.pdf